CLINICAL TRIAL: NCT03703999
Title: Efficacy and Acceptance of Freestyle Libre Abbott Use in Real Life in Type 1 Diabetic Patients
Brief Title: Freestyle Libre Use in Real Life: Efficacy and Acceptance
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Daniela Bruttomesso, MD, PhD, University of Padova
Other Study IDs: 4465/AO/18
Record Dates: First submitted 2018-09-20; First posted 2018-10-12 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: flash glucose monitoring; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- type 1 diabetic patients freestyle Libre: group of type 1 diabetic patients that will be selected to use Freestyle libre on the basis of clinicians decisions and reimbursement criteria
  Interventions: Device: Type 1 diabetic patients freestyle libre

INTERVENTIONS:
Device: Type 1 diabetic patients freestyle libre — patients selected to use freestyle libre

SUMMARY:
Aim of the study is to evaluate efficacy of freestyle Libre system (flash glucose monitoring) in real life in term of Glycated Haemoglobin reduction and acceptance of the system evaluated through validated questionnaires after 3 and 6 months of device's use.

DETAILED DESCRIPTION:
Freestyle Libre is a new technology developed to monitor glycemic values in diabetic patients.

The system is available in Italy from 2014 but in Veneto region reimbursement for insulin treated diabetic patients is available from august 2017.

International trial (for example Impact trial) demonstrated efficacy of the system (reduction of the time spent in hypoglycemia).

Aim of this study is to evaluate efficacy in real life in term of glycated haemoglobin (HbA1c) reduction. The investigators will enrollee in this trial all type 1 diabetic patients that will start to use the system, on the basis of clinicians decisions and reimbursement criteria.

Investigators will evaluate changes in HbA1c and changes in hypoglycameia fear and therapy acceptance through validated questionnaires after 3 and 6 months of system use

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of at least 18 years of age
* Diagnosis of type 1 diabetes mellitus (diagnosed according to World Health Organization criteria) for at least 1 year
* Availability to wear Freestyle Libre sensor
* Signature of informed consent

Exclusion Criteria:

* Pregnancy, breastfeeding, intention to undergo pregnancy
* Known allergies to skin patches or disinfectants used during the study.
* Skin lesions, irritation, redness, edema in sites where sensors can be applied, as this might interfere with sensor's placement
* Use of drugs that may interfere with glucose metabolism (such as steroids) unless they are chronic therapies whose dosage has remained stable over the past 3 months and is expected to remain stable during the study period.
* Severe medical or psychological conditions, which, in the opinion of the medical team, may compromise patients' safety while using freestyle LIbre sensor
* Patients enrolled in other clinical trials.
* patients that usually wear other continuous glucose monitoring system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 1 diabetic patients selected by clinicians to start Freestyle Libre use
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 3 and 6 months
  changes in HbA1c values

SECONDARY OUTCOMES:
changes in hypoglycemia fear | after 3 and 6 months
  Evaluation of hypoglycemia fear through a validated questionnaires, Hypoglycemic Fear Survey (HFS-II). The questionnaires is composed by 33 questions with a Linkert Scale (0-4)
changes in therapy satisfaction | after 3 and 6 months
  Evaluation of changes in therapy satisfaction through a validated questionnaires, Diabetes Treatment Satisfaction Questionnaire (DTSQ). The questionnaires is composed by 8 questions with a Linkert Scale (0-6)
hypoglycemic episodes | after 3 and 6 months
  number of hypoglycemic episodes
weight | after 3 and 6 months
  changes in weight (Kg)
insulin use | after 3 and 6 months
  changes in insulin dose (unit/Kg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No